CLINICAL TRIAL: NCT01708551
Title: Histological Analysis and Correlation With Ultrasound Imaging to Evaluate the Safety and Effectiveness of Treating Axillary Hyperhidrosis Subjects With the Ulthera® System
Brief Title: Histological Analysis Following Ulthera System Treatment for Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-134
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2015-10

CONDITIONS: Hyperhidrosis
Keywords: Hyperhidrosis; Axillary sweating; Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Active Comparator): Subjects naïve to Ultherapy™ for treatment of hyperhidrosis will receive bilateral Ulthera System treatments; dual depth treatment at 4.5mm and 3.0mm.
  Interventions: Device: Ulthera System Treatment
- Group B (Active Comparator): Subjects who were non-responders to a prior Ultherapy™ treatment for hyperhidrosis will receive bilateral Ulthera System treatments; dual depth treatment at 4.5mm and 3.0mm.
  Interventions: Device: Ulthera System Treatment
- Group C (Active Comparator): Subjects will receive one double-density Ulthera System treatment; dual depth treatment at 4.5mm and 3.0mm.
  Interventions: Device: Ulthera System Treatment
- Group D (Active Comparator): Subjects naïve to Ultherapy™ for treatment of hyperhidrosis will receive bilateral Ulthera System treatments at 2.0mm treatment depth and standard energy level.
  Interventions: Device: Ulthera System Treatment
- Group E (Active Comparator): Subjects naïve to Ultherapy™ for treatment of hyperhidrosis will receive bilateral Ulthera System treatments at 2.0mm treatment depth and adjusted energy level.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 60 subjects will be enrolled into one of five treatment groups. Subjects enrolled in Groups A, B or C will undergo axillary punch biopsies during the course of the trial to determine the number and depth of the sweat glands, and receive dual depth treatments (4.5mm and 3.0mm); either two bilateral Ultherapy™ treatments to the axillas 30 days apart (Groups A and B) or one bilateral Ultherapy™ treatment (Group C). Subjects in Groups D and E will receive two bilateral Ultherapy™ treatments to the axillas 30 days apart at a 2.0mm treatment depth and two different energy settings (Group D at 0.45 J, Group E at 0.30 J). Protocol amended (Sept 2014): Subjects in Groups D and E will receive treatments at the same energy setting (0.30J) and two treatment densities: Group D, 60 lines/treatment square; Group E, 40 lines per treatment square. Follow-up visits will occur at 7, 30, 90 and 180 days post-treatment #2.

DETAILED DESCRIPTION:
This study is a prospective, single-center, non-randomized pilot clinical trial. Subjects enrolled will include:

* those naïve to Ultherapy™ for treatment of hyperhidrosis (Group A, n=31); dual-depth treatment at 4.5mm and 3.0mm;
* those who were non-responders to a prior Ultherapy™ treatment for hyperhidrosis (Group B, n=approx 5), dual-depth treatment at 4.5mm and 3.0mm;
* those naïve to Ultherapy™ for treatment of hyperhidrosis who will receive one double-density study treatment (Group C, n=4), dual-depth treatment at 4.5mm and 3.0mm;
* those naïve to Ultherapy™ for treatment of hyperhidrosis (Group D, n=10), single-depth treatment at 2.0mm at standard energy;
* those naïve to Ultherapy™ for treatment of hyperhidrosis (Group E, n=10), single-depth treatment at 2.0mm at adjusted energy.
* Protocol amended (Sept 2014): Subjects in Groups D and E will receive treatments at the same energy setting (0.30J) and two treatment densities: Group D, 60 lines/treatment square; Group E, 40 lines per treatment square.

Ultrasound images will be captured of each axilla to assess dermal thickness and depth of sweat glands. A gravimetric measurement of sweat production and starch iodine test will be performed prior to treatment. Digital images of the starch iodine test will be obtained. Hyperhidrosis Disease Severity Scale (HDSS)scores will be obtained prior to each treatment. During treatment, the average Numeric Rating Scale (NRS) score will be obtained by axilla treated. Efficacy will be determined by a reduction in the number of sweat glands from baseline to 90-days post-treatment, as evidenced by histological analysis. Subject Gravimetric results, Starch iodine results, and HDSS scores at all follow-ups compared to baseline will also be analyzed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18-75
* Subject is in good health
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies
* Groups A, C, D and E: At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature / humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.) Group B: A mean of >50mg/5min of sweat production following a prior Ultherapy treatment.
* A HDSS score is 3 or 4. An attempt will be made to approximate an equal number of scores 3 and 4.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Absence of physical conditions unacceptable to the investigator.
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control.

Exclusion Criteria:

* Dermal disorder including infection at anticipated treatment sites in either axilla.
* Previous botulinum toxin treatment of the axilla in the past year.
* Expected use of botulinum toxin for the treatment of any other disease during the study period.
* Known allergy to starch powder, iodine, lidocaine, or epinephrine.
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Unwillingness to wash off deodorants and abstain use 72 hours prior to treatments or assessments.
* Subjects with a history of a bleeding disorder
* Use of cholinomimetics, anticholinergics, or any oral herbal medicine treatments for hyperhidrosis.
* Inability to withhold use of antiperspirants and deodorants, or any other topical treatments for hyperhidrosis within 72 hours prior to study treatments and assessments.
* Unwillingness for complete shaving or removal of underarm hair within 12 hours prior to study treatments and follow-up visits.
* Women who are pregnant, lactating, possibly pregnant or planning a pregnancy during the study period.
* Inability to understand the protocol or to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of sweat glands from baseline to 90-days post-treatment. | 90 days post-treatment
  Based on histological analyses of biopsied, Ultherapy™-treated, tissue, the changed in the number of sweat glands present at 90days post-treatment will be compared to the number of sweat glands present at baseline.

SECONDARY OUTCOMES:
Reduction in spontaneous axillary sweat production assessed by gravimetric method at 90-days post treatment | 7 days post-treatment
  A 50% reduction or more in Gravimetric measure at 7 days post-treatment compared to baseline.
Reduction in spontaneous axillary sweat production assessed by gravimetric method at 90-days post treatment | 30 days post-treatment
  A 50% reduction or more in Gravimetric measure at 30 days post-treatment compared to baseline.
Reduction in spontaneous axillary sweat production assessed by gravimetric method at 90-days post treatment | 90 days post-treatment
  A 50% reduction or more in Gravimetric measure at 90 days post-treatment compared to baseline.
Reduction in spontaneous axillary sweat production assessed by gravimetric method at 90-days post treatment | 180 days post-treatment
  A 50% reduction or more in Gravimetric measure at 180 days post-treatment compared to baseline.
HDSS score reduction | 90 days post-treatment
  HDSS score reduction from a 3 or 4 to a 1 or 2
Starch iodine test | 90 days post-treatment
  Assess the reduction in starch iodine test area at 90 days post-treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, PhD, Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States